CLINICAL TRIAL: NCT07038616
Title: Observation of the Response to Ovulation Induction on the Day of Intrauterine Insemination and Correlation Between Progesterone Level and Pregnancy Rate (OVUL-IIU)
Brief Title: Observation of the Response to Ovulation Triggering on the Day of Intrauterine Insemination and Correlation Between Progesterone Level and Pregnancy Rate (OVUL-IIU)
Acronym: OVUL-IIU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: OVUL-IIU
Record Dates: First submitted 2025-05-19; First posted 2025-06-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Infertility
Keywords: Stimulated cycle; intrauterine insemination; clinical pregnancy rate; donor sperm; progesterone; ovulation induction; ovulation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intrauterine inseminations (IUI) are a commonly used technique in assisted reproductive technology (ART) to help women conceive, whether within a couple or as single individuals. However, national success rates remain modest, with an average live birth rate of 10% per cycle, which leads many ART centers to favor in vitro fertilization (IVF) as a more effective option.

Nevertheless, IUI retains several advantages: it is less invasive, less expensive, and, when appropriately indicated, can achieve satisfactory outcomes.

Guidelines exist for ovarian stimulation protocols prior to IUI, aimed at optimizing the chances of success. So far, no clear superiority has been demonstrated between pharmacological ovulation triggering and spontaneous ovulation. However, accurate timing of insemination in relation to ovulation is recognized as a key factor for success.

Very few studies have focused on the response to ovulation triggering, and none have explored a correlation with clinical pregnancy rates.

Yet, monitoring of the luteal phase and response to ovulation triggering is a common practice in ART, particularly in the context of frozen embryo transfers (FET), suggesting that these parameters may be worth further investigation in the context of IUI.

Hence, the interest of this study is to determine whether there is a correlation between progesterone levels and clinical pregnancy rates in patients undergoing intrauterine insemination (IUI).

DETAILED DESCRIPTION:
This is a single-center observational cohort study with retrospective and prospective data collection.

Participation in the study is offered in the CHIC MPA department. Data will be collected over a 12-month period.

The research consists of retrieving data from the patient's and spouse's medical records and from software for presenting biological laboratory results .

Patients and their spouses will be informed of the study orally, and will receive a written information note.

ELIGIBILITY:
Inclusion Criteria:

* Single women or couples, heterosexual or homosexual, undergoing insemination at the medically assisted procreation.center
* Aged 18 to 43
* Any indication for IUI in compliance with the Recommendations for Good Practices in MPA (RBP)
* Blood test on the day of insemination with estradiol, progesterone, LH and hCG measured as part of routine care

Exclusion Criteria:

-Opposition of patients to data collection

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of single women or couples, heterosexual or homosexual, undergoing insemination at a medically assisted procreation (MAP) center. Participants are aged between 18 and 43 years old. They have an indication for intrauterine insemination (IUI) in accordance with the Recommendations for Good Practices in Assisted Reproductive Medicine (RBP). . Only those who have had a blood as part of routine care on the day of insemination, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Rate of early pregnancies based on progesterone levels measured on the day of ovulation trigger | 6-7 weeks Gestational Age
  Rate of early pregnancies based on progesterone levels measured on the day of ovulation trigger

SECONDARY OUTCOMES:
Rate of early pregnancies (HCG > 100) and ultrasound (6-7 weeks gestational age) | 6-7 weeks Gestational Age
  Rate of early pregnancies (HCG > 100) and ultrasound (6-7 weeks gestational age)
Rate of spontaneous miscarriage | From enrollment until 12 weeks Gestational Age
  Rate of spontaneous miscarriage before 12 weeks Gestational Age
Estradiol level the morning of the insemination (pg/ml) | The morning of the insemination (between 1 and 4 hours before the insemination)
  Estradiol level will be collected for each patient The morning of the insemination (between 1 and 4 hours before the insemination)
LH level the morning of the insemination (UI/L) | The morning of the insemination (between 1 and 4 hours before the insemination)
  LH level will be collected for each patient , the morning of the insemination (between 1 and 4 hours before the insemination)
hCG level the morning of the insemination (UI/L) | The morning of the insemination (between 1 and 4 hours before the insemination)
  hCG level will be collected for each patient , the morning of the insemination (between 1 and 4 hours before the insemination)and 4 hours before the insemination)
Progesterone level the morning of the insemination (ng/ml) | The morning of the insemination (between 1 and 4 hours before the insemination)
  Progesterone level will be collected for each patient , the morning of the insemination (between 1 and 4 hours before the insemination)
Time between first IUI and early pregnancy (HCG > 100 (UI/L) | From first IUI until HCG > 100 (UI/L)
  Time between first IUI and early pregnancy (HCG > 100 (UI/L)
Predictive factor for pregnancy: BMI ( kg/m^2) | From enrollment until the morning of insemination (between 1 and 4 hours before insemination)
  Predictive factor for pregnancy: BMI
Predictive factor for pregnancy:number of inseminated spermatozoa (millions) | From enrollment until the morning of insemination (between 1 and 4 hours before insemination)
  Predictive factor for pregnancy: number of inseminated spermatozoa
Predictive factor for pregnancy: age (years) | From enrollment until the morning of insemination (between 1 and 4 hours before insemination)
  Predictive factor for pregnancy: age

CONTACTS AND LOCATIONS:
Locations (1):
- Chi Creteil, Créteil, CHI Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided